CLINICAL TRIAL: NCT00841659
Title: Randomized, 2-Way Crossover, Bioequivalence Study of Paroxetine Hydrochloride 40 mg Film-Coated Tablets and Paxil® 40 mg Film-Coated Tablets Administered as 1 x 40 mg Film-Coated Tablet in Healthy Subjects Under Fed Conditions
Brief Title: Paroxetine Hydrochloride 40 mg Tablets Under Fed Conditions
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Teva Pharmaceuticals USA (Industry)
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: 02183-A
Record Dates: First submitted 2009-02-09; First posted 2009-02-11 (Estimated); Results first posted 2009-08-18 (Estimated); Last update posted 2024-08-19 (Actual); Status verified 2024-08

CONDITIONS: Healthy
Keywords: Bioequivalence; Healthy Subjects
MeSH Terms: interventions — Paroxetine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Paroxetine (Experimental): Paroxetine HCl 40 mg Tablet (test) dosed in first period followed by Paxil® 40 mg Tablet (reference) dosed in second period
  Interventions: Drug: Paroxetine HCl
- Paxil® (Active Comparator): Paxil® 40 mg Tablet (reference) dosed in first period followed by Paroxetine HCl 40 mg Tablet (test) dosed in second period
  Interventions: Drug: Paxil®

INTERVENTIONS:
Drug: Paroxetine HCl — 40 mg Film-Coated Tablet
  Arms: Paroxetine
Drug: Paxil® — 40 mg Film-Coated Tablet
  Arms: Paxil®

SUMMARY:
The objective of this study is to compare the rate and extent of absorption of paroxetine hydrochloride 40 mg film-coated tablets (test) and Paxil® (reference) administered as 1 x 40 mg film-coated tablet under fed conditions.

DETAILED DESCRIPTION:
Criteria for Evaluation: FDA Bioequivalence Criteria

Statistical Methods: FDA bioequivalence statistical methods

ELIGIBILITY:
Inclusion Criteria

* Subjects will be females and/or males, non-smokers, 18 years of age and older.
* Female Subjects will be post-menopausal or surgically sterilized.
* Post-menopausal status is defined as absence of menses for the past 12 months,
* Sterile status is defined as hysterectomy, bilateral oophorectomy or tubal ligation at least 6 months ago.

Exclusion Criteria

Subjects to whom any of the following applies will be excluded from the study:

* Clinically significant illnesses within 4 weeks of the administration of study medication.
* Clinically significant surgery within 4 weeks prior to the administration of the study medication.
* Any clinically significant abnormality found during medical screening.
* Subjects with a history of renal, hepatic or cardiovascular disease, tuberculosis, epilepsy, asthma, diabetes, psychosis or glaucoma will not be eligible for this study.
* History or presence of any clinically significant gastrointestinal pathology (e.g. chronic diarrhea, inflammatory bowel diseases), unresolved gastrointestinal symptoms (e.g. diarrhea, vomiting), liver or kidney disease or other conditions known to interfere with the absorption, distribution, metabolism or excretion of the drug.
* Subjects with a history of seizures.
* Subjects who have already had an episode of mania.
* Any reason which, in the opinion of the medical subinvestigator, would prevent the subject from participating in the study.
* Abnormal laboratory tests judged clinically significant.
* Positive urine drug screen at screening.
* Positive testing for hepatitis B, hepatitis C or HIV at screening.
* ECG abnormalities (clinically significant) or vital sign abnormalities (systolic blood pressure lower than 90 or over 140 mmHg, or diastolic blood pressure lower than 50 or over 90; or heart rate less than 50 bpm or over 100 bpm) at screening.
* Subjects with BMI ≥30.0.
* History of significant alcohol abuse within six months of the screening visit or any indication of the regular use of more than two units of alcohol per day (1 Unit = 150 mL of wine or 360 mL of beer or 45 mL of alcohol 40%).
* History of drug abuse or use of illegal drugs: use of soft drugs (such as marijuana) within 3 months of the screening visit or hard drugs (such as cocaine, phencyclidine (PCP) and crack) within 1 year of the screening visit.
* Any food allergy, intolerance, restriction or special diet that, in the opinion of the medical subinvestigator, contraindicates the subject's participation in this study.
* History of allergic reactions to paroxetine hydrochloride or other related drugs (e.g. citalopram hydrobromide, fluoxetine hydrochloride, fluvoxamine maleate and sertraline hydrochloride).
* History of allergic reactions to heparin.
* Use of any drugs known to induce or inhibit hepatic drug metabolism (examples of inducers: barbiturates, carbamazepine, phenytoin, glucocorticoids, rifampin/rifabutin; examples of inhibitors: antidepressants, cimetidine, diltiazem, erythromycin, ketoconazole, MAO inhibitors, neuroleptics, verapamil, quinidine, valproic acid, use of an investigational drug or participation on an investigation study within 30 days prior to the administration of the study medication.
* Use of prescription medication within 14 days prior to administration of study medication or over-the-counter products )including natural products, vitamins, garlic as a supplement) within 7 days prior to administration of study medication, except for topical products without systemic absorption.
* Subjects who have had a depot injection or an implant of any drug 3 months prior to administration of study medication.
* Donation of plasma (500 mL) within 7 days. Donation or loss of whole blood prior to administration of the study medication as follows:
* Less than 300 mL of whole blood within 30 days or
* 300 mL to 500 mL of whole blood within 45 days or
* more than 500 mL of whole blood within 56 days.
* Positive alcohol breath test at screening.
* Subjects who have used tobacco in any form within the 90 days preceding study drug administration.
* Intolerance to venipuncture.

Additional exclusion criteria for female subjects only:

* Breast feeding subjects.
* Positive urine pregnancy test at screening (performed on all females).

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2002-08; Primary Completion 2002-08 (Actual); Study Completion 2002-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Benoit Girard, MD, Principal Investigator — Anapharm
Locations (1):
- Anapharm Inc., Sainte-Foy, Quebec, Canada

RESULTS

PARTICIPANT FLOW:
Groups:
- Paroxetine (Test) First: Paroxetine HCl 40 mg Tablet (test) dosed in first period followed by Paxil® 40 mg Tablet (reference) dosed in second period
- Paxil® (Reference) First: Paxil® 40 mg Tablet (reference) dosed in first period followed by Paroxetine HCl 40 mg Tablet (test) dosed in second period
Period: First Intervention
Arm/Group | Paroxetine (Test) First | Paxil® (Reference) First
Started | 12 | 12
Completed | 12 | 12
Not Completed | 0 | 0
Period: Washout: 2 Weeks
Arm/Group | Paroxetine (Test) First | Paxil® (Reference) First
Started | 12 | 12
Completed | 11 | 12
Not Completed | 1 | 0
Not completed — Protocol Violation | 1 | 0
Period: Second Intervention
Arm/Group | Paroxetine (Test) First | Paxil® (Reference) First
Started | 11 | 12
Completed | 11 | 12
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Paroxetine (Test) First | Paxil® (Reference) First | Total
Number analyzed (Participants) | 12 | 12 | 24
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 12 | 12 | 24
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 2 | 3
  Male | 11 | 10 | 21
Race/Ethnicity, Customized [Number; unit: Participants]
  Caucasian | 11 | 12 | 23
  Asian | 1 | 0 | 1
Region of Enrollment [Number; unit: participants]
  Canada | 12 | 12 | 24

OUTCOME MEASURES:

1. Primary Outcome: Cmax - Maximum Observed Concentration (of Paroxetine in Plasma)
Description: Bioequivalence based on Cmax
Time Frame: Blood samples collected over 120 hour period
Population: Data from all subjects who completed the study were included in the statistical analysis.
Measure: Mean (Standard Deviation); unit: ng/mL
Groups:
- Paroxetine: Paroxetine HCl 40 mg Tablet (test) dosed in either period
- Paxil®: Paxil® 40 mg Tablet (reference) dosed in either period
Arm/Group | Paroxetine | Paxil®
Number analyzed (Participants) | 23 | 23
ng/mL | 24.66 (13.25) | 24.22 (12.51)
Statistical Analysis 1: Comparison: Paroxetine vs Paxil®; Test type: Non-Inferiority or Equivalence — Using GLM procedures in SAS, analysis of variance (ANOVA)was performed on log-transformed AUC0-t, AUC0-inf and Cmax at the significance level of 0.05; Ratio of LS Means x 100 = 99.96 — Bioequivalence is established when ratio of means falls within 80-125

2. Primary Outcome: AUC0-inf - Area Under the Concentration-time Curve From Time Zero to Infinity (Extrapolated)
Description: Bioequivalence based on AUC0-inf
Time Frame: Blood samples collected over 120 hour period
Population: Data from all subjects who completed the study were included in the statistical analysis.
Measure: Mean (Standard Deviation); unit: ng*h/mL
Arm/Group | Paroxetine | Paxil®
Number analyzed (Participants) | 23 | 23
ng*h/mL | 797.53 (830.95) | 873.69 (974.14)
Statistical Analysis 1: Comparison: Paroxetine vs Paxil®; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; Ratio of LS Means x 100 = 93.58 — Bioequivalence is established when ratio of means falls within 80-125

3. Primary Outcome: AUC0-t - Area Under the Concentration-time Curve From Time Zero to Time of Last Non-zero Concentration (Per Participant)
Description: Bioequivalence based on AUC0-t
Time Frame: Blood samples collected over 120 hour period
Population: Data from all subjects who completed the study were included in the statistical analysis.
Measure: Mean (Standard Deviation); unit: ng*h/mL
Arm/Group | Paroxetine | Paxil®
Number analyzed (Participants) | 23 | 23
ng*h/mL | 741.41 (685.80) | 787.19 (736.20)
Statistical Analysis 1: Comparison: Paroxetine vs Paxil®; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; Ratio of LS Means x 100 = 94.29 — Bioequivalence is established when ratio of means falls within 80-125

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Principal Investigator is not permitted to discuss or publish trial results.